CLINICAL TRIAL: NCT05243212
Title: A Phase 1/2, Open-Label, Dose Escalation and Confirmation Study of CAR-BCMA, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against BCMA in Subjects With Multiple Myeloma
Brief Title: Study of CAR-BCMA, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against BCMA in Subjects With Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Hila Magen, Head of Multiple Myeloma Unit in Sheba Medical Center, Sheba Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-21-8048-HM-CTIL
Record Dates: First submitted 2021-10-11; First posted 2022-02-16 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma; Relapse Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: The treatment dose is 6 or 9 x 10^6 CAR+ T cells/kg of recipient bodyweight.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'low' dose (Experimental): The dose escalation stage will involve recruitment of 3 RRMM patients for 'low' dose (6 x 106 CAR-T cells/kg) CAR-T therapy. After 14 days of follow-up for each of the 3 subjects, the DSC will determine whether the next subject can be recruited. After 14 days follow-up for the 3rd subject, DSC will review data for the 3rd subject and consider the data for the first 3 subjects.
  Interventions: Biological: CAR-BCMA
- 'high' dose (Experimental): In the absence of dose limiting toxicities (DLTs), the DSC may recommend recruitment of 3 subjects to be treated with the 'high' dose (9x106 CAR-T cells/kg) CAR-T therapy, with similar staggering.
  Interventions: Biological: CAR-BCMA

INTERVENTIONS:
Biological: CAR-BCMA — CAR-BCMA T-cells are genetically modified autologous T-cells directed to the B-cell maturation antigen (BCMA). CAR-BCMA T-cells identify and eliminate BCMA-expressing malignant plasma cells. Upon binding to BCMA-expressing cells, the CAR transmits a signal to promote T cell expansion, activation, persistence and elimination of malignant plasma cells.

SUMMARY:
This is an open label, abbreviated (3+3) dose escalation study in subjects with RRMM, followed by an extension phase at the selected safe dose. The dose escalation stage will involve recruitment of 3 RRMM patients for 'low' dose (6 x 106 CAR-T cells/kg) CAR-T therapy. After 14 days of follow-up for each of the 3 subjects, the DSC will determine whether the next subject can be recruited.

After 14 days follow-up for the 3rd subject, DSC will review data for the 3rd subject and consider the data for the first 3 subjects. In the absence of dose limiting toxicities (DLTs), the DSC may recommend recruitment of 3 subjects to be treated with the 'high' dose (9x106 CAR-T cells/kg) CAR-T therapy, with similar staggering. In case of DLTs in one of the 3 low dose subjects, the DSC may recommend to recruit an additional 3 low dose subjects (6 in total). If there are no additional DLTs in these 3 patients the low dose may be recommended by the DSC for the extension stage. However, further DLTs may prompt the DSC to recommend to modify the protocol, or to stop the study. In case of DLTs in one of the first 3 high dose subjects, the DSC may recommend to recruit an additional 3 high dose subjects.If there are no additional DLTs in these 3 patients, the high dose may be recommended by the DSC for the study extension stage. However, further DLTs may prompt the DSC to recommend continuation to the extension stage with the low dose, or to modify the protocol, or to stop the study.

After completion of two months follow-up for the 6th subject in the low or high dose cohort (as applicable), and review of all the data for all subjects, following DSC recommendations, the Stage 2 extension phase of the study may recruit additional subjects, up to a maximum of 75 subjects for Stages 1 and 2, combined.

DSC will review study data during the extension stage follow-up after 5 years to determine if additional safety follow-up is required.

ELIGIBILITY:
Inclusion Criteria:

1. Bone marrow plasma cells must be at least 10% of total bone marrow cells based on a bone marrow biopsy/aspiration performed within 30 days of the start of protocol treatment.
2. Documented diagnosis of multiple myeloma according to IMWG diagnostic criteria.
3. Subjects must have measurable MM as defined by at least one of the criteria below.

   One or more of these abnormalities defines measurable disease
   1. Serum M-protein equal or greater than 0.4 g/dl (10 g/l).
   2. Urine M-protein equal or greater than 200 mg/24 h.
   3. Serum free light chain (FLC) assay: involved FLC level greater or equal to10 mg/dl (100 mg/l) provided serum FLC ratio is abnormal.
   4. A biopsy-proven plasmacytoma
4. Patients must have received at least 3 prior treatment regimens for multiple myeloma.
5. Greater than or equal to 18 years of age.
6. Able to understand and sign the Informed Consent Document.
7. Clinical performance status of ECOG 0-2
8. Subjects of both genders must be willing to practice birth control from the time of enrollment on this study and for four months after receiving the preparative regimen.
9. Women of child bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
10. Seronegative for HIV- 1, 2 antibody.
11. Seronegative for hepatitis B surface antigen (HBsAg) or HBsAg positive with negative PCR for HBV nucleotides in blood. (Treatment to prevent HBV reactivation is standard in any case of seropositivity for HBV).
12. Seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then subjects must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
13. Syphilis negative.
14. Absolute neutrophil count greater than or equal to 500/mm3 without the support of filgrastim or other growth factors.
15. Platelet count greater than or equal to 30,000/mm3 without transfusion support
16. Hemoglobin greater than 8.0 g/dl.
17. Less than 5% plasma cells in the peripheral blood leukocytes
18. At least 14 days must have elapsed since any prior systemic therapy at the time the subject starts the cyclophosphamide and fludarabine conditioning regimen, and subjects' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
19. Systemic anti-myeloma therapy including systemic corticosteroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to the required leukapheresis, within 2 weeks prior to CAR T-cell infusion, and for 30 days after the CAR T cell infusion, unless required for treatment of toxicity or other medical need.
20. Cardiac ejection fraction greater than or equal to 45% by echocardiography within 6 weeks of the start of the treatment protocol.

Exclusion Criteria:

1. Subjects with second malignancies in addition to multiple myeloma are not eligible if the second malignancy has required treatment within the past 3 years or is not in complete remission. There are two exceptions to this criterion: successfully treated non-metastatic basal cell or squamous cell skin carcinoma.
2. Women who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
3. Active systemic infections (defined as infections causing fevers or requiring antimicrobial treatment), or other major uncontrolled medical illnesses.
4. Active HBV and HCV infection which is identified by positive PCR to viral nucleotides in blood.
5. Systemic corticosteroid steroid therapy of greater than 5 mg/day of prednisone or equivalent dose of another corticosteroid are not allowed within 2 weeks prior to either the required leukapheresis or the initiation of the conditioning chemotherapy regimen.
6. Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN) and direct bilirubin > 2 x ULN
7. Inadequate renal function defined by serum creatinine clearance /estimated clearance of ≤ 20(ml/min).
8. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
9. Subjects with CNS involvement.
10. Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 15 days prior to leukapheresis for CAR T-cell manufacture, or is currently enrolled in an investigational study. However, prior therapy with belantamab mafotodin can be used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-09-19 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 2 months
  Overall response rate, two months after CAR-BCMA T-cell infusion determined in accordance with the International Myeloma Working Group (IMWG) guidance.
CAR BCMA related toxicity | 2 years
  Frequency of CAR-BCMA related toxicities: CRS and ICANS, according to ASTCT consensus grading (Lee 2019).
CAR BCMA related toxicity | 2 years
  Any AEs according to common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
progression free survival | 12 months
  PFS is defined as the time CAR T -cell infusion to the date of either first documented relapse, progression or death due to any cause.
overalll free survival | 12 months
  OS was defined as the time from CART-cell infusion to death of any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel